CLINICAL TRIAL: NCT07311564
Title: A Phase 2, Randomized, Placebo-controlled, Double-blind Clinical Study to Evaluate Efficacy and Safety of LAD603 in Adult Subjects With Severe to Very Severe Alopecia Areata
Brief Title: A Study of LAD603 in Adults With Alopecia Areata
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M-00223-20; 2025-523342-27-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-29; First posted 2025-12-31 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Alopecia Areata
Keywords: Hair Loss; Hypotrichosis; Alopecia
MeSH Terms: conditions — Alopecia Areata; Alopecia; Hypotrichosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LAD603 Dose A (Experimental): Participants will receive LAD603 Dose A , Subcutaneous (SC) injection from Day 1 up to 28 weeks.
  Interventions: Drug: LAD603
- LAD603 Dose B (Experimental): Participants will receive LAD603 Dose B, SC injection from Day 1 up to 28 weeks.
  Interventions: Drug: LAD603
- LAD603 Dose C (Experimental): Participants will receive LAD603 Dose C, SC injection from Day 1 up to 28 weeks.
  Interventions: Drug: LAD603
- Placebo for LAD603 (Placebo Comparator): Participants will receive Placebo for LAD603 SC injection from Day 1 up to 28 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LAD603 — LAD603 administered subcutaneously.
  Arms: LAD603 Dose A; LAD603 Dose B; LAD603 Dose C
Other: Placebo — LAD603 matching placebo administered subcutaneously.
  Arms: Placebo for LAD603

SUMMARY:
The main aim of the study is to evaluate the effect of LAD603 in adult participants with severe to very severe alopecia areata (AA). The study will also evaluate the safety, pharmacokinetics (PK), immunogenicity and pharmacodynamic (PD) biomarkers of LAD603.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female between 18 and 65 years old at the time of signing the informed consent.
* Severe to very severe AA criteria:

  1. Greater than or equal to (>=) 50% hair loss of the scalp as measured by SALT without evidence of terminal hair regrowth within 6 months at both the Screening and Baseline (Day 1) visits.
  2. Current episode of hair loss lasting at least 6 months and not exceeding 7 years.
* Participants who are WOCBP or male must agree to the requirements for the avoidance of pregnancy and exposure of the participant's partner to LAD603 during the study,

Exclusion Criteria:

AA, Skin Specific, and Other Inflammatory Diseases

* Participants have other types of alopecia (including but not limited to traction, scarring alopecia).
* Participants with "diffuse" type AA.
* Currently has an active form of other inflammatory skin disease(s) or evidence of skin condition (e.g., psoriasis, seborrheic dermatitis, lupus) at the time of the Screening or Baseline (Day 1) visits that is expected to interfere with the assessment of alopecia areata severity.

Other Medical Conditions

* Participant has previous severe adverse reaction to subcutaneously administered medication.
* Participant has any of the following liver safety laboratory results at Screening

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than or equal to (>=) 2.5 × upper limit of normal (ULN)
  2. Total bilirubin (TBL) >=1.5 × ULN (TBL >=3 × ULN in participants with Gilbert's syndrome)
  3. Alkaline phosphatase (ALP) >=1.5 × ULN

     Prior/Concomitant Therapy
* Intention to use any concomitant medication that is not permitted by this protocol or failure to undergo the required washout period for a particular prohibited medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-05-23 (Estimated); Study Completion 2027-11-21 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in the Severity of Alopecia Tool (SALT) Score | Baseline, Week 28
  The SALT score is the sum of percentage of hair loss in all areas with a maximum score of 100 (higher score indicates greater hair loss).

SECONDARY OUTCOMES:
Percentage of Participants Achieving an Absolute SALT Score Less than or Equal to (<=) 10/20 | At Week 28
  Percentage of participants achieving an absolute SALT score of <= 10/20. The SALT score is the sum of percentage of hair loss in all areas with a maximum score of 100 (higher score indicates greater hair loss). Total percentage of patients with absolute SALT score of <= 10/20 will be calculated.
Percentage of Participants Achieving a Clinician-Reported Outcome (ClinRO) for Eyelash Hair Loss of 0/1 | At Week 28
  The ClinROs for Eyelash Hair Loss is a clinician reported assessment which measures the severity and impact of hair loss in these specific areas. It comprises a 4-point category response options (0 to 3) rating the extent of eyebrow hair loss. This scale ranges from no hair loss (0) to complete hair loss (3).
Percentage of Participants Achieving a ClinRO for Eyebrow Hair Loss of 0/1 | At Week 28
  The ClinROs for Eyebrow Hair is a clinician reported assessment which measures the severity and impact of hair loss in these specific areas. It comprises a 4-point category response options (0 to 3) rating the extent of eyebrow hair loss. This scale ranges from no hair loss (0) to complete hair loss (3).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.
Locations (1):
- Investigator Site 1, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No